CLINICAL TRIAL: NCT04050618
Title: Multi-Center Cross-Over Evaluation Of Avaira Vitality Silicone Hydrogel Contact Lens and Two Hydrogel Lenses in Daily Wear
Brief Title: Evaluation Of One Silicone Hydrogel Contact Lens and Two Hydrogel Lenses in Daily Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-103
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be masked to lens type. Investigators will be unmasked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ocufilcon D control lens, then fanfilcon A test lens (Experimental): Participants will wear the ocufilcon D control lens for 4 weeks, then crossover to fanfilcon A test lens for 4 weeks of daily wear.
  Interventions: Device: fanfilcon A test lens; Device: ocufilcon D control lens
- etafilcon A controls, then fanfilcon A test lens (Experimental): Participants will wear the etafilcon D control lens for 2 weeks, then crossover to fanfilcon A test lens for 2 weeks of daily wear.
  Interventions: Device: fanfilcon A test lens; Device: etafilcon A control lens

INTERVENTIONS:
Device: fanfilcon A test lens — Silicone hydrogel contact lens
  Other Names: test lens; Avaira Vitality
Device: ocufilcon D control lens — hydrogel contact lens
  Other Names: Biomedics 55 Premier; ocufilcon D (4-weekly) control lens
  Arms: ocufilcon D control lens, then fanfilcon A test lens
Device: etafilcon A control lens — hydrogel contact lens
  Other Names: etafilcon A (2-weekly) control lens; Acuvue 2
  Arms: etafilcon A controls, then fanfilcon A test lens

SUMMARY:
To evaluate the comparative clinical performance of the fanfilcon A silicone hydrogel lens used in daily wear and to compare this with competitive hydrogel lens products.

DETAILED DESCRIPTION:
This 8-week, subject-masked, bilateral, two-part, cross-over evaluation will compare the clinical performance of fanfilcon A silicone hydrogel contact lens and competitive hydrogel contact lenses when worn daily. Lenses will be replaced either on a 2-weekly or 4-weekly basis, depending on control lens group.

ELIGIBILITY:
Inclusion Criteria:

* Be a currently adapted soft contact lens wearer (>1 month of lens wear).
* Be at least 18 years of age.
* Refractive astigmatism <1.00D in both eyes.
* Have clear corneas and be free of any anterior segment disorders.
* Be correctable through spherocylindrical refraction to 20/25 or better in each eye.
* Contact lens sphere requirement between -1.00D and -6.00D (inclusive).
* Require visual correction in both eyes (monovision allowed, no monofit).
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:

  1. No amblyopia
  2. No strabismus
  3. No evidence of lid abnormality or infection
  4. No conjunctival abnormality or infection that would contraindicate contact lens wear
  5. No clinically significant slit lamp findings (i.e. corneal staining, stromal edema, staining, scarring, vascularization, infiltrates or abnormal opacities)
  6. No other active ocular disease.
* Own a mobile phone and be able to respond to SMS survey during the period 8am-8pm.
* Willing to comply with the wear and study visit schedule.

Exclusion Criteria:

* Using CooperVision Avaira Vitality, J&J Acuvue 2 or CooperVision Biomedics 55.
* Require toric or multifocal contact lenses.
* Previously shown a sensitivity to any of the study solution components.
* Any systemic or ocular disease or allergies affecting ocular health.
* Using systemic or topical medications that will in the investigator's opinion affect ocular physiology or lens performance.
* Clinically significant (>Grade 3) corneal staining, corneal stromal edema, corneal vascularization, tarsal abnormalities, bulbar hyperemia, limbal hyperemia, or any other abnormality of the cornea that would contraindicate contact lens wear.
* Any corneal infiltrates or any corneal scarring or neovascularization within the central 5mm of the cornea.
* Keratoconus or other corneal irregularity.
* Aphakia or amblyopia.
* Have undergone corneal refractive surgery or any anterior segment surgery.
* Abnormal lacrimal secretions.
* Has diabetes.
* Known/reported infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV).
* History of chronic eye disease (e.g. glaucoma).
* Pregnant or lactating or planning a pregnancy at the time of enrolment.
* Participation in any concurrent clinical trial or in last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-06-09 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Ardaya, OD, Principal Investigator — Golden Optometric Group; William J Bogus, OD, Principal Investigator — Office of William J. Bogus, O.D.; Bryan E Frazier, OD, Principal Investigator — Frazier Vision, Inc; Wayne Golden, OD, Principal Investigator — Golden Vision; Andrew J Sacco, OD, Principal Investigator — Sacco Eye Group; Christopher Pearson, OD, Principal Investigator — Omega Vision Center PA (DBA Sabal Eye Care)
Locations (6):
- United States (6):
  - Golden Optometric Group, Whittier, California
  - Omega Vision Center PA (DBA Sabal Eye Care), Longwood, Florida
  - Golden Vision, Sarasota, Florida
  - Sacco Eye Group, Vestal, New York
  - Frazier Vision, Inc, Tyler, Texas
  - Office of William J. Bogus, O.D., Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | Ocufilcon D Control Lens, Then Fanfilcon A Test Lens | Etafilcon A Controls, Then Fanfilcon A Test Lens
Started | 58 | 56
Completed | 56 | 56
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Second Intervention
Arm/Group | Ocufilcon D Control Lens, Then Fanfilcon A Test Lens | Etafilcon A Controls, Then Fanfilcon A Test Lens
Started | 56 | 56
Completed | 55 | 56
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocufilcon D Control Lens, Then Fanfilcon A Test Lens | Etafilcon A Controls, Then Fanfilcon A Test Lens | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 56 | 114
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (9.42) | 32.7 (9.00) | 33.1 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 41 | 79
  Male | 20 | 15 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 46 | 45 | 91
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 56 | 52 | 108
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 56 | 114

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Comfort Rating
Description: Subjective overall comfort rating was assessed on a 0-10 subjective scale, 0=extremely uncomfortable, 10=can't feel lenses
Time Frame: Two weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ocufilcon D - Group A: Subjects were randomized to wear ocufilcon D control lens for four weeks.
  Ocufilcon D - hydrogel contact lens
- Fanfilcon A - Group A: Subjects were randomized to wear fanfilcon A test lens for four weeks.
  Fanfilcon A - SiHy contact lens
- Etafilcon A - Group B: Subjects were randomized to wear etafilcon A control lens for two weeks.
  Etafilcon A - hydrogel contact lens
- Fanfilcon A - Group B: Subjects were randomized to wear fanfilcon A test lens for two weeks.
  Fanfilcon A - SiHy contact lens
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
units on a scale | 8.2 (2.04) | 8.6 (1.19) | 8.3 (1.72) | 8.3 (1.64)

2. Primary Outcome: Subjective Overall Comfort Rating
Description: as for outcome 1
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
units on a scale | 7.9 (2.10) | 8.6 (1.26)

3. Secondary Outcome: Average Wearing Time
Description: Average wearing time - measured by time of day using 24-hour clock, to the nearest 10 minutes
Time Frame: Two weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
hours/day | 14.01 (1.689) | 14.7 (1.674) | 13.84 (1.756) | 13.80 (1.757)

4. Secondary Outcome: Average Wearing Time
Description: Average wearing time - measured by time of day using 24-hour clock, to the nearest 10 minutes
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
hours/day | 14.21 (1.501) | 14.42 (1.504)

5. Secondary Outcome: Average Comfortable Wearing Time
Description: Average comfortable wearing time was assessed by time of day when first aware of lenses using 24-hour clock, to the nearest 10 minutes.
Time Frame: Two weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
hours/day | 11.60 (3.743) | 12.45 (3.669) | 12.18 (3.210) | 11.67 (3.330)

6. Secondary Outcome: Average Comfortable Wearing Time
Description: as for outcome 5
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
hours/day | 11.37 (3.869) | 12.40 (3.379)

7. Secondary Outcome: Lens Centration
Description: Lens centration will be recorded in the scale of 0 to 2 (0=centered - optimal, 1 = decentered slightly, 2 = substantially decentered (>0.5mm)).
Time Frame: Baseline (after 15 minutes)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 58 | 56 | 56 | 56
Number analyzed (eyes) | 116 | 112 | 112 | 112
percentage of eyes
  Optimal | 85 | 93 | 91 | 94
  Slight | 15 | 7 | 9 | 6
  Substantial | 0 | 0 | 0 | 0

8. Secondary Outcome: Lens Centration
Description: as for outcome 7
Time Frame: Two weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
Number analyzed (eyes) | 114 | 112 | 112 | 112
percentage of eyes
  Optimal | 88 | 93 | 83 | 95
  Slight | 12 | 7 | 17 | 5
  Substantial | 0 | 0 | 0 | 0

9. Secondary Outcome: Lens Centration
Description: as for outcome 7
Time Frame: Four weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
Number analyzed (eyes) | 112 | 110
percentage of eyes
  Optimal | 86 | 89
  Slight | 14 | 11
  Substantial | 0 | 0

10. Secondary Outcome: Corneal Coverage
Description: Corneal coverage (yes=full corneal coverage all times / no=incomplete corneal coverage)
Time Frame: Baseline (after 15 minutes of lens dispense)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 58 | 56 | 56 | 56
Number analyzed (eyes) | 116 | 112 | 112 | 112
percentage of eyes
  yes | 100 | 100 | 100 | 100
  no | 0 | 0 | 0 | 0

11. Secondary Outcome: Corneal Coverage
Description: Corneal coverage (yes=full corneal coverage all times / no=incomplete corneal coverage)
Time Frame: Two weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
Number analyzed (eyes) | 114 | 112 | 112 | 112
percentage of eyes
  yes | 98 | 98 | 100 | 100
  no | 2 | 2 | 0 | 0

12. Secondary Outcome: Corneal Coverage
Description: Corneal coverage (yes=full corneal coverage all times / no=incomplete corneal coverage)
Time Frame: Four weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
Number analyzed (eyes) | 112 | 110
percentage of eyes
  yes | 100 | 98
  no | 0 | 2

13. Secondary Outcome: Post-Blink Movement
Description: Post-blink movement measured by scale 0-4 (0=insufficient, 1=minimal, unacceptable movement, 2=optimal movement, 3=moderate, but acceptable movement, 4=excessive, unacceptable movement)
Time Frame: Baseline (after 15 minutes of lens dispense)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 58 | 56 | 56 | 56
Number analyzed (eyes) | 116 | 112 | 112 | 112
percentage of eyes
  Insufficient | 0 | 0 | 2 | 0
  Minimal | 4 | 0 | 9 | 5
  Optimal | 91 | 94 | 84 | 82
  Moderate | 5 | 6 | 5 | 13
  Excessive | 0 | 0 | 0 | 0

14. Secondary Outcome: Post-Blink Movement
Description: as for outcome 13
Time Frame: Two weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
Number analyzed (eyes) | 114 | 112 | 112 | 112
percentage of eyes
  Insufficient | 0 | 0 | 0 | 0
  Minimal | 4 | 0 | 11 | 5
  Optimal | 91 | 98 | 83 | 91
  Moderate | 5 | 2 | 6 | 4
  Excessive | 0 | 0 | 0 | 0

15. Secondary Outcome: Post-Blink Movement
Description: as for outcome 13
Time Frame: Four weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
Number analyzed (eyes) | 112 | 110
percentage of eyes
  Insufficient | 0 | 0
  Minimal | 4 | 2
  Optimal | 80 | 96
  Moderate | 16 | 2
  Excessive | 0 | 0

16. Secondary Outcome: Lens Tightness - Push-up Test
Description: Lens tightness - push-up test 0-100% continuous scale (100%=movement, 50%=optimum, 0%=Falls from cornea without lid support)
Time Frame: Baseline (after 15 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 58 | 56 | 56 | 56
Number analyzed (eyes) | 116 | 112 | 112 | 112
percentage of eyes | 49.6 (5.36) | 49.0 (3.80) | 52.1 (8.26) | 50.2 (5.69)

17. Secondary Outcome: Lens Tightness - Push-up Test
Description: as for outcome 16
Time Frame: Two weeks
Measure: Mean (Standard Deviation); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
Number analyzed (eyes) | 114 | 112 | 112 | 112
percentage of eyes | 49.7 (4.12) | 48.4 (4.55) | 50.6 (5.88) | 48.0 (7.95)

18. Secondary Outcome: Lens Tightness - Push-up Test
Description: as for outcome 16
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
Number analyzed (eyes) | 112 | 110
percentage of eyes | 48.4 (5.62) | 49.8 (3.67)

19. Secondary Outcome: Overall Lens Fit Acceptance
Description: Overall lens fit acceptance - Graded on a scale of 0-4 (0=should not be worn, 1=borderline but not acceptable, 2=minimal acceptable, 3=not perfect but OK to dispense, 4=perfect)
Time Frame: Baseline (after 15 minutes of lens dispense)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 58 | 56 | 56 | 56
Number analyzed (eyes) | 116 | 112 | 112 | 112
percentage of eyes
  Should not be worn | 0 | 0 | 0 | 0
  Borderline | 0 | 0 | 0 | 0
  Minimal | 0 | 0 | 0 | 0
  OK | 22 | 9 | 18 | 21
  Perfect | 78 | 91 | 82 | 79

20. Secondary Outcome: Overall Lens Fit Acceptance
Description: as for outcome 19
Time Frame: Two weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
Number analyzed (eyes) | 114 | 112 | 112 | 112
percentage of eyes
  Should not be worn | 0 | 0 | 0 | 0
  Borderline | 0 | 0 | 0 | 0
  Minimal | 0 | 0 | 0 | 0
  OK | 16 | 12 | 26 | 13
  Perfect | 84 | 88 | 74 | 88

21. Secondary Outcome: Overall Lens Fit Acceptance
Description: as for outcome 19
Time Frame: Four weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
Number analyzed (eyes) | 112 | 110
percentage of eyes
  Should not be worn | 0 | 0
  Borderline | 0 | 0
  Minimal | 0 | 0
  OK | 23 | 15
  Perfect | 77 | 85

22. Secondary Outcome: Rating of Lens Surface Wettability
Description: Lens surface wettability rated on the appearance on the lens surface (0-4 scale, 0=Very poor: immediately displaying non-wetting areas on lens surface, 4=Excellent: appearance of a healthy cornea with very long drying time).
Time Frame: Baseline (after 15 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 58 | 56 | 56 | 56
Number analyzed (eyes) | 116 | 112 | 112 | 112
units on a scale | 3.93 (0.266) | 3.96 (0.172) | 3.94 (0.286) | 3.92 (0.265)

23. Secondary Outcome: Rating of Lens Surface Wettability
Description: as for outcome 22
Time Frame: Two weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
Number analyzed (eyes) | 114 | 112 | 112 | 112
units on a scale | 3.74 (0.490) | 3.69 (0.512) | 3.73 (0.611) | 3.80 (0.437)

24. Secondary Outcome: Rating of Lens Surface Wettability
Description: as for outcome 22
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
Number analyzed (eyes) | 112 | 110
units on a scale | 3.55 (0.736) | 3.81 (0.365)

25. Secondary Outcome: Presence of Film Deposits
Description: Presence of film deposits on front surface of the lens graded 0-4 (0=No film, 1=Slight film visible only under magnification, 2=Moderate film only under magnification, 3=Moderate film visible to the naked eye, 4=heavy film visible to the naked eye).
Time Frame: Two weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
Number analyzed (eyes) | 114 | 112 | 112 | 112
percentage of eyes
  Grade 0 | 85 | 86 | 85 | 86
  Grade 1 | 12 | 13 | 13 | 13
  Grade 2 | 3 | 2 | 2 | 2
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 1 | 0

26. Secondary Outcome: Presence of Film Deposits
Description: as for outcome 25
Time Frame: Four weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
Number analyzed (eyes) | 112 | 110
percentage of eyes
  Grade 0 | 74 | 79
  Grade 1 | 22 | 17
  Grade 2 | 2 | 2
  Grade 3 | 0 | 0
  Grade 4 | 2 | 2

27. Secondary Outcome: Number of White Spot Deposits
Description: Number of white spot deposits assessed using slit lamp with white light, low medium magnification
Time Frame: Two weeks
Measure: Mean (Standard Deviation); unit: number of white spots
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
Number analyzed (eyes) | 114 | 112 | 112 | 112
number of white spots | 0.01 (0.094) | 0.05 (0.567) | 0.03 (0.211) | 0.22 (1.145)

28. Secondary Outcome: Number of White Spot Deposits
Description: Number of white spot deposits assessed using slit lamp with white light, low medium magnification
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: number of white spots
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
Number analyzed (eyes) | 112 | 110
number of white spots | 0.15 (0.988) | 0.18 (0.940)

29. Secondary Outcome: Primary Gaze Lag
Description: Primary gaze lag measured by scale 0-4 (0=insufficient, 1=minimal, unacceptable movement, 2=optimal movement, 3=moderate, but acceptable movement, 4=excessive, unacceptable movement)
Time Frame: Baseline (after 15 minutes of lens dispense)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 58 | 56 | 56 | 56
Number analyzed (eyes) | 116 | 112 | 112 | 112
eyes
  Insufficient | 0 | 0 | 2 | 0
  Minimal | 5 | 0 | 8 | 6
  Optimal | 107 | 106 | 100 | 93
  Moderate | 4 | 6 | 2 | 13
  Excessive | 0 | 0 | 0 | 0

30. Secondary Outcome: Primary Gaze Lag
Description: as for outcome 29
Time Frame: Two weeks
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
Number analyzed (Participants) | 57 | 56 | 56 | 56
Number analyzed (eyes) | 114 | 112 | 112 | 112
eyes
  Insufficient | 0 | 0 | 0 | 0
  Minimal | 2 | 0 | 8 | 2
  Optimal | 108 | 109 | 97 | 108
  Moderate | 4 | 3 | 7 | 2
  Excessive | 0 | 0 | 0 | 0

31. Secondary Outcome: Primary Gaze Lag
Description: as for outcome 29
Time Frame: Four weeks
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 56 | 55
Number analyzed (eyes) | 112 | 110
eyes
  Insufficient | 0 | 0
  Minimal | 2 | 2
  Optimal | 96 | 106
  Moderate | 14 | 2
  Excessive | 0 | 0

32. Secondary Outcome: Comfort Throughout the Day
Description: Comfort throughout the day was assessed on a scale of 0-10 (0=extremely uncomfortable, 10=cannot feel the lenses) using text message responses
Time Frame: Day 3 - 8:00am
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fanfilcon A - Group A: Subjects were randomized to wear fanfilcon A test lens for four weeks.
  fanfilcon A - SiHy contact lenses
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 43 | 45
units on a scale | 8.55 (1.607) | 9.22 (1.146)

33. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 3 - 12:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 52 | 48
units on a scale | 8.58 (1.601) | 9.27 (1.180)

34. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 3 - 4:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 48 | 48
units on a scale | 8.85 (1.384) | 8.71 (1.458)

35. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 3 - 8:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 55 | 46
units on a scale | 8.11 (1.912) | 8.57 (1.377)

36. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 7 - 8:00am
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 40 | 44
units on a scale | 8.13 (1.727) | 8.84 (1.328)

37. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 7 - 12:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 48 | 43
units on a scale | 8.48 (1.750) | 8.98 (1.336)

38. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 7 - 4:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 49 | 45
units on a scale | 8.39 (1.869) | 8.84 (1.261)

39. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 7 - 8:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 50 | 45
units on a scale | 8.22 (1.920) | 8.48 (1.722)

40. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 12 - 8:00am
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 47 | 39
units on a scale | 8.28 (1.896) | 8.85 (1.348)

41. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 12 - 12:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 47 | 51
units on a scale | 8.68 (1.721) | 8.73 (1.387)

42. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 12 - 4:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 50 | 50
units on a scale | 8.34 (1.710) | 8.56 (1.459)

43. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 12 - 8:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 51 | 49
units on a scale | 8.22 (2.023) | 8.39 (1.382)

44. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 26 - 8:00am
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 40 | 43
units on a scale | 8.35 (1.861) | 8.58 (1.277)

45. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 26 - 12:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 50 | 45
units on a scale | 8.22 (1.741) | 8.80 (1.392)

46. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 26 - 4:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 51 | 47
units on a scale | 8.04 (1.876) | 8.62 (1.609)

47. Secondary Outcome: Comfort Throughout the Day
Description: as for outcome 32
Time Frame: Day 26 - 8:00pm
Population: Overall number of participants analyzed differ based on the number of text responses received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A
Number analyzed (Participants) | 52 | 48
units on a scale | 7.79 (2.127) | 8.29 (1.774)

ADVERSE EVENTS:
Time Frame: From dispense up to 4 weeks for ocufilcon D and fanfilcon A - Group A, from dispense up to 2 weeks for etafilcon A and fanfilcon A - Group B. A total of 8 weeks
Arm/Group | Ocufilcon D - Group A | Fanfilcon A - Group A | Etafilcon A - Group B | Fanfilcon A - Group B
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57 | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57 | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 2/58 | 0/57 | 0/56 | 0/56
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocufilcon D - Group A (N=58) | Fanfilcon A - Group A (N=57) | Etafilcon A - Group B (N=56) | Fanfilcon A - Group B (N=56)
headache (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04050618/Prot_SAP_000.pdf